CLINICAL TRIAL: NCT05287789
Title: Effectiveness of Squatting Position on Constipation Severity and Defecation Problems in the Postoperative Period of Hernia Surgery
Brief Title: Effectiveness of Squatting Position on Constipation Severity and Defecation Problems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meltem Kaya (Other)
Responsible Party: Sponsor-Investigator, Meltem Kaya, Lecturer, MSc, Karabuk University
Organization: Karabuk University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SQUATTING; KBYBAB-17/YL-454 (Other Grant/Funding Number: Karabuk University Scientific Research Projects Office)
Record Dates: First submitted 2021-03-18; First posted 2022-03-18 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Constipation; Postoperative Care; Nursing Care
Keywords: Squatting Position; Constipation; Defecation problems; Clinical Nursing Research
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Intervention Model Description: pretest-posttest time series model with the different control group
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Squatting position by footstool (Experimental): After the first postoperative ambulation, stable patients whose bowel movements resumed met their initial defecation needs with the squatting position created using a footstool at the appropriate height on the water closet type toilet.
  The patients used footstools in the hospital and throughout a week after discharge at home for defecation.
  Interventions: Other: Squatting position by footstool
- Control Group (No Intervention): The control group received the routine care provided to all the patients in the clinic with no additional interventions.

INTERVENTIONS:
Other: Squatting position by footstool — Before the study, the height of the toilet bowls in the patient rooms was measured as 42 cm. The stools to be used for the study are manufactured by ordering laminated with white medium density fiberboard and synthetic resin resistant to harsh chemicals. Stools are made of high quality non-slip materials for patient safety.
  After the first postoperative ambulation, stable patients whose bowel movements resumed met their initial defecation needs with the squatting position created using a stool at the appropriate height on the water closet type toilet.
  The patients used footstools throughout a week after discharge at home and in the hospital for defecation.
  Arms: Squatting position by footstool

SUMMARY:
One of the most common nursing care problems after surgery is defecation problems and the risk of constipation. The aim of the study was to determine the effectiveness of the squatting position with footstool on the constipation severity and defecation problems in the postoperative period in patients with hernia surgery.

DETAILED DESCRIPTION:
In this study, after the surgical procedure, the patients were placed in a squatting position by placing a stool under their feet in the toilet.

ELIGIBILITY:
Inclusion Criteria:

* Hernia surgery in the general surgery clinic
* Between 18 and 65 years of age
* BMI between normal and overweight (18.50-24,99 kg/m2: Normal,25-29,99 kg/m2: Overweight)
* Being able to establish verbal communication
* Volunteering to participate in the study
* Absence of mental confusion
* Having full consciousness and orientation
* Having no communication difficulties
* Having a constipation risk between moderate to high
* Using a water closet type toilet at home

Exclusion Criteria:

* Having a low risk of constipation
* Patient who declined to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Change from before surgery in The Constipation Severity Scale (CSS) average score | Data were collected before surgery, post-op 1st day, post-op 2nd day and on the 7th day after discharge. All of the patients were discharged on the 2nd postoperative day.
  Constipation Severity Scale (CSS) aims to determine individuals' defecation frequency, intensity, and difficulty. The CSS consists of 16 items and three sub dimensions, namely Excrement Congestion, Large Bowel Laziness, and Pain. The lowest score that can be attained from the CSS is 0 while the highest score that can be attained is 73.

SECONDARY OUTCOMES:
Difficulty pushing in defecation average score | Data were collected post-op 2nd day and on the 7th day after discharge. All of the patients were discharged on the 2nd postoperative day.
  Average score on a scale from 0 to 4. 0 I did not experience any difficulties, 1 I had mild difficulties, 2 I had some difficulties, 3 I had a lot of difficulties, 4 I experienced extreme difficulties.
Duration of defecation, average minutes | Data were collected post-op 2nd day and on the 7th day after discharge. All of the patients were discharged on the 2nd postoperative day.
  The time (minutes) the patient spent defecation.
Defecation pain average score | Data were collected post-op 2nd day and on the 7th day after discharge. All of the patients were discharged on the 2nd postoperative day.
  The Visual Analog Scale (VAS) consists of a 10 cm line used to evaluate defecation pain by scoring it between 1 and 10.
Stool consistency | Data were collected post-op 2nd day and on the 7th day after discharge. All of the patients were discharged on the 2nd postoperative day.
  Bristol Stool Scale (BSS) is designed to classify the form of human faeces into seven categories. Types 1-2, hard; types 3-5, normal; types 6-7, loose/liquid
Fear of pushing in defecation average score | Data were collected post-op 2nd day and on the 7th day after discharge. All of the patients were discharged on the 2nd postoperative day.
  Average score on a scale from 0 to 4. 0 No Fear, 1 Slightly Scared, 2 Slightly Scared, 3 Very Afraid, 4 Extremely Too Afraid.

CONTACTS AND LOCATIONS:
Overall Officials: Meltem Kaya, Principal Investigator — Karabuk University; Aysegul Oksay Sahin, Study Chair — Karabuk University; Isıl Isık Andsoy, Study Chair — Karabuk University
Locations (1):
- Karabuk University, Karabük, Turkey (Türkiye)